CLINICAL TRIAL: NCT03862573
Title: A Pragmatic Randomized Controlled Trial of Virtual Reality vs. Standard-of-Care for Comfort During Dental Treatment
Brief Title: Virtual Reality vs. Standard-of-Care for Comfort During Dental Procedures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ran Goldman, Professor and Co-head of the Division of Clinical Pharmacology, Division of Emergency Medicine, Department of Pediatrics; Investigator, BC Children's Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H19-00486
Record Dates: First submitted 2019-03-02; First posted 2019-03-05 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Dental Procedures
Keywords: Virtual Reality; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants are distracted by wearing the virtual reality headset and watching a roller coaster app during the dental procedure
  Interventions: Device: Virtual Reality
- Control (Standard of Care) (No Intervention): Participants are distracted with Standard-of-Care by dentists and/or parents.

INTERVENTIONS:
Device: Virtual Reality — Participants wear a Virtual Reality headset that consists of a ASUS phone and a VOX+ Z3 3D Virtual Reality Headset. The phone runs the VR Roller Coaster app to produce the virtual environment.
  Arms: Virtual Reality

SUMMARY:
Children sometimes need dental procedures which can be painful and associated with child pain and anxiety. In addition to pain medication, distraction may help children cope with the pain. This may include interacting with books, TV, toys or videogames.

Virtual Reality (VR) is an immersive experience using sight, sound, and position sense. Using VR may enhance distraction during the painful procedure and may reduce attention to pain.

This study will randomize children (4 - 16 years old) to receive Virtual Reality or standard of care in addition to local anesthetics during dental procedures. Pain, anxiety and satisfaction will be measured as well as the amount of analgesics used and the timing of the procedure. Outcome measures will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Children age 4 to < 17 years
2. Arriving to the UBC dentistry clinic and need dental assessment/procedures
3. Parents will sign a consent form and children will sign an assent form

Exclusion Criteria:

1. Children with conditions that may prohibit participation or evaluation of the procedure (such as developmental delay, autism, challenging communication)
2. Facial features prohibiting wearing the VR goggles
3. Children needing sedation that includes inhalation via a mask (N2O) or IV/IM sedation

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2019-03-31 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Post Procedure Pain using the Faces Pain Scale - Revised | Pain is reported by children immediately following completion of the procedure (within two minutes post-procedure). This scale should take less than one minute to complete
  Level of pain as reported by children using Faces Pain Scale - Revised. The scale includes six faces that represent progressively more intense features of pain. Children point to the face that best represents their current level of pain. The minimum score is 0 (representing least pain) and the maximum score is 10 (representing greater pain). The scale increase in increments of 2.

SECONDARY OUTCOMES:
Post Local Anesthetic Pain using the Faces Pain Scale - Revised | Pain is reported by children immediately following injection of the local anesthetic (within two minutes post-injection). This scale should take less than one minute to complete
  Level of pain as reported by children using Faces Pain Scale - Revised. The scale includes six faces that represent progressively more intense features of pain. Children point to the face that best represents their current level of pain. The minimum score is 0 (representing least pain) and the maximum score is 10 (representing greater pain). The scale increase in increments of 2.
Anxiety using the Venham Situational Anxiety Score | Anxiety is reported by children immediately following completion of the procedure (within two minutes post-procedure). This scale should take less than one minute to complete
  Level of Situational Anxiety as reported by children using the Venham Situational Anxiety Score. This scale includes 8 sets of 2 images of children which represent differing levels of anxiety. Children point to the child that best represents them in that instance. In each set of 2 images of children, one represents greater anxiety (scored as 1) and one represents lesser anxiety (scored as 0). The points from each set of images are totaled. The minimum score is 0 (least anxious) and maximum score is 8 (most anxious).
Co-operation of the child as measured by the Dentist on 100mm VAS | Co-operation is rated immediately following completion of the dental visit.
  The dentist will rate their impression of the level of co-operation by the child on a 100 mm VAS.
Patient Satisfaction determined qualitatively by an open ended question | Satisfaction question is reported by children immediately following completion of the dental procedure
  Satisfaction from the procedure is determined qualitatively. Children are asked "What is your opinion on how the procedure went?" Answers will be recorded in writing and be assessed for themes (similar words, positive or negative language).
Parent Satisfaction determined qualitatively by an open ended question | Satisfaction question is reported by parents immediately following completion of the dental procedure
  Satisfaction from the procedure is determined qualitatively. Parents are asked "What is your opinion on how the procedure went?" Answers will be recorded in writing and be assessed for themes (similar words, positive or negative language).

CONTACTS AND LOCATIONS:
Locations (1):
- UBC graduate pediatric dentistry clinic, Vancouver, British Columbia, Canada